CLINICAL TRIAL: NCT03911167
Title: An Analysis of Clinical Efficacy Based on the Robotic, Laparoscopic, and Open Approach in Radical Resection of Rectal Cancer
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2019LSK-009
Record Dates: First submitted 2019-03-26; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-01

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Laparoscopy; Robotics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- RG: RG: robotic group
  Interventions: Procedure: open, laparoscopic, and robotic
- LG: LG:laparoscopic group,
  Interventions: Procedure: open, laparoscopic, and robotic
- OG: OG：open group
  Interventions: Procedure: open, laparoscopic, and robotic

INTERVENTIONS:
Procedure: open, laparoscopic, and robotic — Radical resection of rectal cancer in robotic, laparoscopic, and open approach

SUMMARY:
A retrospective study was done on the medical records for 24 rectal cancer patients underwent robotic proctectomy from September 2017 to July 2018 at the First Afﬁliated Hospital of Xi'an Jiaotong University.In the same department,a total of 25 patients who treated with laparoscopic proctectomy and 24 patients underwent open proctectomy were were selected as controls in a 1:1:1 ratio. Comparing the perioperative conditions and hospitalization related costs of the three groups.

ELIGIBILITY:
Inclusion Criteria:

* endoscopic biopsy pathological diagnosis of rectal cancer is clear, preoperative CT, MRI examination did not see the tumor directly invaded the surrounding organs;
* blood test, cardiac ultrasound, lung ventilation function and other preoperative examination without absolute surgical contraindications;
* without distant metastasis such as liver, lung, bone, and abdominal cavity.

Exclusion Criteria:

* there is distant organ transfer or extensive abdominal metastasis;
* emergency surgery for acute intestinal obstruction, hemorrhage, perforation, intestinal rupture, etc.;
* combined with other primary malignant tumors;
* other colonectomy and combined with other organ resection;
* patients with severe basic diseases unable to tolerate surgery;
* pregnant and lactating women;
* patients who underwent neoadjuvant radiotherapy and chemotherapy before surgery;
* those who underwent palliative surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Postoperative complication rate，% | 2 weeks

SECONDARY OUTCOMES:
Urine tube time,days; | 2 weeks
operation time,minutes; | 2 weeks
intraoperative bleeding,ml; | 2 weeks
number of lymph node detection, | 2 weeks
exhaust time,days; | 2 weeks
intake time, days; | 2 weeks
postoperative hospital stay,days; | 2 weeks
hospitalization expenses,yuan | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No